CLINICAL TRIAL: NCT04461418
Title: An Interventional, Randomized Phase II Study Investigating the Efficacy of Immune Checkpoint Inhibitors While Corticosteroid Therapy is Required for Patients With Symptomatic Brain Metastases.
Brief Title: Accelerated Checkpoint Therapy for Any Steroid Dependent Patient With Brain Metastases
Acronym: ACT-FAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0003
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, two cohort, permuted block randomization phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Dose starting at 4 mg daily (for patients randomized to the Dexamethasone arm).
  Interventions: Drug: Glucocorticoid therapy
- Prednisone (Active Comparator): Dose starting at 25 mg/day (a calculation of equipotent steroid equivalencies will be used).
  Interventions: Drug: Glucocorticoid therapy

INTERVENTIONS:
Drug: Glucocorticoid therapy — The study intervention is defined as treatment with either prednisone or dexamethasone as palliative therapy for the control of neurological symptoms; patients with symptomatic brain metastases with a requirement for glucocorticoid therapy will be treated with an available, standard-of-care immune checkpoint inhibitor regimen.

SUMMARY:
Immunotherapy treatments are intended to boost a person's immune system to fight their cancer. Treatment with immunotherapy has been shown to be effective in a wide range of cancers, including melanoma skin cancer, lung cancer and kidney cancer, among others.

Steroids are anti-inflammatory medications which may suppress the immune system. For this reason, persons requiring treatment with steroids have not previously been allowed to participate in immunotherapy clinical trials. Therefore, we do not know whether or not immunotherapy treatments are effective in patients who are also receiving treatment with steroids.

When cancer has spread to the brain swelling may occur around the tumors, and headache, nausea, seizures or stroke-like symptoms may occur. In this instance, steroids are important to reduce swelling within the brain, thus alleviating these symptoms.

Because patients requiring treatment with steroids have not previously been allowed to participate in immunotherapy clinical trials, we do not know whether treatment with immunotherapy is effective when steroid treatments are also used. This study will investigate this question, and also attempt to determine whether treatment with one steroid versus another results in a better response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the following histologically confirmed diagnoses will be eligible for enrolment: malignant melanoma, non-small cell lung cancer and renal cell carcinoma and genitourinary carcinoma not-otherwise specified.
2. At the time of enrolment patients must have central nervous system metastases requiring corticosteroid therapy and have already started corticosteroid therapy.
3. Patients eligible for treatment with an available, standard-of-care immune checkpoint inhibitor regimen.
4. Patients with extracranial disease will be eligible for enrolment, however the presence of extracranial measurable disease is not a requirement for enrolment.
5. Patients must be 18 years of age or older.
6. Patients must be capable of providing consent to enrolment and willing to comply with study treatment and follow-up.
7. Patients with a performance status of ECOG 0-2 will be eligible for enrolment.
8. Measurable intracranial disease must be present according to RECIST 1.1 criteria.
9. Patients with hyperthyroidism or hypothyroidism but that are stable on hormone replacement will not be excluded.
10. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
11. Patients of childbearing / reproductive potential should use adequate birth control methods, as defined by the investigator, during the study treatment period and for a period of 30 days after the last dose of study drug.
12. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
13. The following adequate organ function laboratory values must be met:

Hematological:

* Absolute neutrophil count (ANC) >1.0
* Platelet count >100
* Hemoglobin >90 mg/dL

Renal:

- Serum creatinine <2x ULN

Hepatic:

* Total serum bilirubin <1.5x ULN
* AST and ALT <3x ULN

Coagulation:

* International Normalized Ratio (INR) <1.5x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Activated Partial Thromboplastin Time (aPTT) <1.5x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)

Exclusion Criteria:

1. Known history of human immunodeficiency virus (HIV), active Hepatitis B or Hepatitis C. Testing for HIV, HBV or HCV is not mandatory for enrolment to study, but may occur at the discretion of the investigator.
2. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
3. Patients receiving non-steroid immunosuppressive agents (examples may include anti-TNF biologic agents, methotrexate, mycophenylate mofetil, tacrolimus) will be excluded from this study.
4. Known prior severe hypersensitivity to study drugs or any component in its formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Intracranial and extracranial objective response rate | 24 weeks following enrolment of the last participant to study
  Objective response rate will be determined utilizing RECIST 1.1 criteria. Baseline staging diagnostic imaging (CT and/or MRI studies) will be performed in advance of beginning treatment and repeated 6 weeks following treatment initiation and at 12 week intervals thereafter.
Time to initiation of therapy | 24 weeks following enrolment of the last participant to study
  Defined as the time interval between first radiographic documentation of intracranial metastatic disease and initiation of systemic immunotherapy.

SECONDARY OUTCOMES:
Mortality analyses | Upon completion of 12 month follow-up period for the final participant enrolled to the study.
  Secondary study outcomes include progression-free and overall survival (PFS, OS). PFS is defined as the time between the date of treatment initiation and the date of disease progression (determined utilizing RECIST 1.1 criteria) or death (whatever the cause), whichever occurs first. For participants who remain alive and whose disease has not progressed, PFS will be censored on the date of last visit/contact with disease assessments. PFS will be based on the disease assessment or date of death provided by the investigator. OS is defined as the time between the date of treatment initiation and the date of death (whatever the cause). For participants who remain alive OS will be censored on the date of last visit/contact with disease assessments. OS will be based on the date of death provided by the investigator.
Patient-reported quality of life analysis | Upon completion of 12 month follow-up period for the final participant enrolled to the study.
  An analysis of patient-reported quality of life will be conducted utilizing the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the EORTC Brain Cancer Module (EORTC QLQ-BN20) questionnaires). Quality of life questionnaires will be administered to participants following enrolment to study but prior to initiation of immunotherapy. Follow-up questionnaires will be administered as part of the standard of care immunotherapy pre-treatment starting 6 weeks from Cycle 1 and every 6 weeks thereafter until end of treatment. Quality of life questionnaires should be administered prior to investigator assessment at each indicated time-point.
Assessment of treatment safety | Upon completion of 12 month follow-up period for the final participant enrolled to the study.
  The Common Terminology Criteria for Adverse Events (CTCAE, version 4.03) will be used to categorize treatment related and non-treatment related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada